CLINICAL TRIAL: NCT05399017
Title: Open-labeled, Non-randomized, Self-controlled Study to Evaluate the Safety and Performance of EZVent in Hospitalized Mechanically Ventilated Patients
Brief Title: Clinical Evaluation of EZVent in Hospitalized Mechanically Ventilated Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Triclinium Clinical Development Middle East and North Africa (Other)
Collaborators: ezz medical Industries (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MD-004
Record Dates: First submitted 2022-05-24; First posted 2022-06-01 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Respiratory Failure; Respiratory Disease
Keywords: EZVent; Ventilator; Mechanical Ventilator; Respiratory failure; medical device; ventilator performance; Egyptian ventilator; ventilator clinical evaluation; ventilator clinical investigation; EZVent clinical evaluation
MeSH Terms: conditions — Respiratory Insufficiency; Respiration Disorders

STUDY DESIGN:
Intervention Model Description: Non-randomized, open-labeled, self-control study, single arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EZVent (Experimental): * Subjects who are involved in the clinical trial are already mechanically ventilated on traditional standard commercial ventilator. Baseline measurements (T0) will be taken from each patient before being transferred to EZVent ventilator. The following measurements will be taken: Vital Signs and hemodynamics (heart rate, blood pressure, temperature, Respiratory rate), Chest X-ray, Arterial blood gases as well as the ventilator mode parameters (dependent on each mode) and lung mechanics parameters (Peak, Plateau, Mean Airway Pressure, Tidal Volume, Airway Resistance and Static Compliance).
  * After taking the baseline measurements, subjects will be disconnected from their traditional standard ventilator and immediately connected to EZVent using the same previous original setting.
  * After 60 & 120 minutes of ventilation on EZVent (T1&T2) respectively, the same measurement will be taken (Vital signs and Hemodynamics will be continuously monitored and recorded every five minutes).
  Interventions: Device: EZVent

INTERVENTIONS:
Device: EZVent — EZVent Ventilator System is designed for respiratory support in hospitalized mechanical ventilated patients. The Ventilator is designed to be used for adults patients. It is designed to be a stationary product suitable for service in hospitals, critical care situations to provide continuous positive pres- sure respiratory support to the patient. The ventilator met EDA, ISO 80601-2-12 requirements on essential performance of critical care ventilator and other applicable international standards.
  Other Names: EZVent Ventilator System

SUMMARY:
Investigation Device: EZVent Ventilator System is designed for respiratory support in hospitalized mechanical ventilated patients. The Ventilator is designed to be used for adults patients. It is designed to be a stationary product suitable for service in hospitals, critical care situations to provide continuous positive pressure respiratory support to the patient. The ventilator met EDA, ISO 80601-2-12 requirements on essential performance of critical care ventilator and other applicable international standards.

Study Title: Open-labeled, non-randomized, self-controlled study to evaluate the safety and performance of EZVent in hospitalized mechanically ventilated patients. Investigational Device EZVent Ventilator System.

Purpose: Evaluation of the safety and performance of EZVent in hospitalized mechanically ventilated patients.

Objectives: Evaluation of the safety and performance of EZVent through monitoring the vital signs and arterial blood gases (ABG) in comparison to a commercial ventilator.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged 18 years or above.
* Mechanically ventilated Patients (on either VC, PC or CPAP modes).
* Able (in the Investigators opinion) and willing to comply with all study requirements.
* Considered clinically stable, with FiO2 less than 60% and PEEP no greater than 10 cm H2O

Exclusion Criteria:

* Pregnant Women
* Patients who experienced myocardial infarction within the last 6 weeks.
* Shocked patients, Hemodynamic instability requiring vasopressors, cardiac arrhythmias, terminal malignancy.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2022-08-15 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Comparable gas exchange parameters | 0-120 minutes
  Comparable gas exchange parameters (PaCO2) at T2 (120 minutes after the patient was on EZVent) in relation to readings at T0 (Baseline readings when the patient was connected to his/ her original standard traditional mechanical ventilator).
Comparable gas exchange parameters | 0-120 minutes
  Comparable gas exchange parameters ( Blood pH values) at T2 (120 minutes after the patient was on EZVent) in relation to readings at T0 (Baseline readings when the patient was connected to his/ her original standard traditional mechanical ventilator)
Comparable gas exchange parameters | 0-120 minutes
  Comparable gas exchange parameters (PaO2) at T2 (120 minutes after the patient was on EZVent) in relation to readings at T0 (Baseline readings when the patient was connected to his/ her original standard traditional mechanical ventilator)
Comparable gas exchange parameters | 0-120 minutes
  Comparable gas exchange parameters (SaO2) at T2 (120 minutes after the patient was on EZVent) in relation to readings at T0 (Baseline readings when the patient was connected to his/ her original standard traditional mechanical ventilator)
Comparable hemodynamic and vital parameters | 0-120 minutes
  Comparable hemodynamic and vital parameters (Blood pressure) at T2 when the patient is on EZVent in relation to at T0
Comparable hemodynamic and vital parameters | 0-120 minutes
  Comparable hemodynamic and vital parameters (pulse) at T2 when the patient is on EZVent in relation to at T0
Comparable hemodynamic and vital parameters | 0-120 minutes
  Comparable hemodynamic and vital parameters (Temperature) at T2 when the patient is on EZVent in relation to at T0
Comparable hemodynamic and vital parameters | 0-120 minutes
  Comparable hemodynamic and vital parameters (Respiratory rate) at T2 when the patient is on EZVent in relation to at T0
Comparable lung mechanics parameters | 0-120 minutes
  Comparable lung mechanics parameters (Static Compliance) at T2 when patient was on EZVent in relation to readings at T0
Comparable lung mechanics parameters | 0-120 minutes
  Comparable lung mechanics parameters (Airway resistance) at T2 when patient was on EZVent in relation to readings at T0
Comparable lung mechanics parameters | 0-120 minutes
  Comparable lung mechanics parameters (Tidal volume) at T2 when patient was on EZVent in relation to readings at T0
Comparable lung mechanics parameters | 0-120 minutes
  Comparable lung mechanics parameters (Mean Airway Pressure) at T2 when patient was on EZVent in relation to readings at T0
Comparable lung mechanics parameters | 0-120 minutes
  Comparable lung mechanics parameters (Plateau) at T2 when patient was on EZVent in relation to readings at T0
Comparable lung mechanics parameters | 0-120 minutes
  Comparable lung mechanics parameters (Peak) at T2 when patient was on EZVent in relation to readings at T0

SECONDARY OUTCOMES:
Serious adverse events | 0-120 minutes
  Serious adverse events (cardiac arrest, pneumothorax, Cardiac tamponade or any other serious medical event)

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Nassar, Prof.Dr, Principal Investigator — Kasr El Aini Hospital
Locations (1):
- Critical Care Unit of Kasr Al-Ainy Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No